CLINICAL TRIAL: NCT03398980
Title: Late Sequelae of Childhood and Adolescent Nasopharyngeal Carcinoma Survivors After Radiotherapy
Status: Completed | Type: Observational
Sponsor: Yuan-hong Gao (Other)
Responsible Party: Sponsor-Investigator, Yuan-hong Gao, Deputy Director，MD & PhD, Professor，Department of Radiation Oncology, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: NPC-C-2017
Record Dates: First submitted 2017-12-29; First posted 2018-01-16 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Childhood and Adolescent; Survivors; Radiotherapy; Late Sequelae
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- survivors treated with CRT: Childhood and Adolescent Nasopharyngeal Carcinoma survivors who were treated with convention radiotherapy (CRT).
  Interventions: Radiation: survivors treated with CRT
- survivors treated with IMRT: Childhood and Adolescent Nasopharyngeal Carcinoma survivors who were treated with intensity-modulated radiotherapy (IMRT).
  Interventions: Radiation: survivors treated with CRT

INTERVENTIONS:
Radiation: survivors treated with CRT — Radiotherapy technology included conventional radiotherapy (CRT) and intensity-modulated radiotherapy (IMRT).
  Other Names: survivors treated with IMRT

SUMMARY:
Although children and adolescents are more likely to have advanced disease at onset, they generally have a significantly better chance of survival. With combined chemotherapy and radiotherapy, overall survival has been reported more than 75% in most pediatric studies. However, little research focuses on long-term morbidities of children and adolescent nasopharyngeal carcinoma (NPC) survivors, and most studies are small scale and have short follow-up time. Therefore, this study analyzed the long-term morbidities of children and adolescent NPC survivors after radiotherapy. Factors associated with those morbidities were also analyzed.

We reviewed the medical records of all NPC patients younger than 18 years old treated at Sun Yat-sen University Cancer Center (SYSUCC) from February 1991 to October 2010. Detailed medical records were taken from our institutional database. Patients were also followed using comprehensive questionnaires and phone calls. We extracted data on clinical characteristics, histopathology, imaging findings, treatment, outcomes, and late morbidities.

Patients with early-stage (stage I and II) disease were treated with radiotherapy alone, and patients with advanced-stage disease (stage III and IV) were treated with a combination of radiotherapy and chemotherapy. Radiotherapy technology included conventional radiotherapy (CRT) and intensity-modulated radiotherapy (IMRT).

We retrospectively reviewed these medical records to collect the required data. All survivors returned to the hospital for follow-up examinations at least every 3 months for the first year, at least every 6 months in the 2nd year, and at least every one year thereafter until the latest follow-up. As part of our routine clinical practice, all patients underwent follow-up MRI examinations of the nasopharynx and neck at least every 6 to 12 months.

Radioactive toxicity on organs was evaluated based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 3.0.

Analyses were performed using SPSS software, version 16.0 (SPSS, Chicago, IL). Chi-squared tests and binary regression analysis were used to compare the CI of treatment comorbidities between different groups of survivors. A P value of 0.05 was chosen as the criteria for statistical significance.

DETAILED DESCRIPTION:
Introduction Nasopharyngeal carcinoma (NPC) is an uncommon childhood malignancy. As the high incidence of local-regional advanced disease, its undifferentiated histology and its close association with Epstein-Barr virus (EBV) , it is distinguishable from the adult form of the disease. Treatment strategies for childhood NPC follow guidelines established for adults. Although children and adolescents are more likely to have advanced disease at onset, they generally have a significantly better chance of survival. With combined chemotherapy and radiotherapy, overall survival has been reported more than 75% in most pediatric studies. However, late sequelae such as endocrinopathies, hearing disorder, dental problems, life-long dry mouth, and secondary neoplasms have been reported. Little research focuses on long-term morbidities of children and adolescent NPC survivors, and most studies are small scale and have short follow-up time. Therefore, this study analyzed the long-term morbidities of children and adolescent NPC survivors after radiotherapy. Factors associated with those morbidities were also analyzed.

Methods and Materials Patients We reviewed the medical records of all NPC patients younger than 18 years old treated at Sun Yat-sen University Cancer Center (SYSUCC) from February 1991 to October 2010. Detailed medical records were taken from our institutional database. Patients were also followed using comprehensive questionnaires and phone calls. All patients were restaged according to the Union for International Cancer Control (UICC) TNM classification version 2009 of NPC. We extracted data on clinical characteristics, histopathology, imaging findings, treatment, outcomes, and late morbidities. Informed consent was obtained from all patients.

Treatment protocols The main treatment strategy for patients was based on the National Comprehensive Cancer Network Guidelines. Patients with early-stage (stage I and II) disease were treated with radiotherapy alone, and patients with advanced-stage disease (stage III and IV) were treated with a combination of radiotherapy and chemotherapy. NPC patients were treated with a high-dose of radiotherapy to the nasopharynx and the involved lymph nodes of the neck, and a moderate dose of radiation to uninvolved nodes and surrounding tissues. Radiotherapy technology included conventional radiotherapy (CRT) and intensity-modulated radiotherapy (IMRT). Patients between 1991 and 2004 received CRT. Post 2004, IMRT became the standard strategy treatment. During the study period, chemotherapy guidelines for NPC were implemented as follows: no chemotherapy for patients with stage I to II disease, and concurrent chemoradiotherapy + neoadjuvant chemotherapy for stage III to IVa-c.

Follow up We retrospectively reviewed these medical records to collect the required data. All survivors returned to the hospital for follow-up examinations at least every 3 months for the first year, at least every 6 months in the 2nd year, and at least every one year thereafter until the latest follow-up. As part of our routine clinical practice, all patients underwent follow-up MRI examinations of the nasopharynx and neck at least every 6 to 12 months.

Evaluation Criterion Radioactive toxicity on organs was evaluated based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 3.0.

Statistical analysis Analyses were performed using SPSS software, version 16.0 (SPSS, Chicago, IL). Chi-squared tests and binary regression analysis were used to compare the CI of treatment comorbidities between different groups of survivors. A P value of 0.05 was chosen as the criteria for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of nasopharyngeal carcinoma.
2. Nasopharyngeal carcinoma patients younger than 18 years old.
3. Nasopharyngeal carcinoma patients who have survived.

Exclusion Criteria:

1. Patients have other diseases.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All NPC patients younger than 18 years old treated at SYSUCC from February 1991 to October 2010.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2016-09-02 (Actual); Primary Completion 2017-01-10 (Actual); Study Completion 2017-01-10 (Actual)

PRIMARY OUTCOMES:
The frequency of some sequelae between survivors treated with CRT and IMRT | up to almost 27 years
  Chi-squared tests and binary regression analysis were used to compare the CI of treatment comorbidities between different groups of survivors. Radioactive toxicity on organs was evaluated based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 3.0.